CLINICAL TRIAL: NCT06011915
Title: A Retrospective Study of Treatment Patterns and Clinical Outcomes in Patients With Central Nervous System Tuberculosis
Status: Completed | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Qin Ning, Director and Chair of Department of Infectious Diseases, Tongji Hospital
Other Study IDs: RETUBO-N
Record Dates: First submitted 2023-08-14; First posted 2023-08-25 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Central Nervous System Tuberculosis
MeSH Terms: conditions — Tuberculosis, Central Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
This is a retrospective clinical study to analyze the clinical characteristics, complications, and effects of different treatment options on long-term prognosis in patients with central nervous system tuberculosis. All cases of central nervous system tuberculosis diagnosed between 2016 and 2021 were included in the electronic medical record system of one center, and data such as demographics, hospitalization information, clinical information, laboratory or imaging examinations, treatment plans, and outcomes were collected.

ELIGIBILITY:
Inclusion Criteria:

* The patient meets the following criteria 1) or 2) or 3):

  1. The discharge diagnosis is central nervous system tuberculosis, refer to the ICD-10 code related to central nervous system tuberculosis.
  2. The discharge diagnosis was tuberculous meningitis (ICD-10: A17.000), or tuberculous cerebrospinal meningitis (ICD-10: A17.001), or tuberculous meningoencephalitis (ICD-10: A17.803 ), or tuberculous encephalitis (ICD-10: A17.804), or tuberculous brain abscess (ICD-10: A17.805), or spinal tuberculosis (ICD-10: A17.806), or tuberculous encephalitis Water (ICD-10: A17.807).
  3. Tuberculous meningitis diagnosed according to the "Guidelines for Diagnosis and Treatment of Central Nervous System Tuberculosis in China (2019 Edition)"
* Age and gender are not limited.

Exclusion Criteria:

* Patients with no clear diagnosis at discharge.
* Patients judged by the investigator to be unsuitable for inclusion in this protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Central nervous system tuberculosis patients came from Wuhan Pulmonary Hospital, which is a third-class A-level specialized hospital integrating tuberculosis prevention and control, clinical diagnosis and treatment of pulmonary diseases, science, teaching and research, located in Wuhan, Hubei Province, China.
Sampling Method: Probability Sample
Enrollment: 638 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
2-year survival rate | 1 years,2 years
  Calculate the 1-year survival rate and 2-year survival rate.
2-year disability rate | 1 years,2 years
  Calculate the 1-year disability rate and 2-year disability rate. Common disabilities include aphasia, hemiplegia, paraplegia, deafness, blindness, mental retardation, etc. For reference, please refer to the 《Grading of Human Injury and Disability Degree》 and 《Guidance for determination of cause-and-effect relationship between personal injury and disease》.

SECONDARY OUTCOMES:
Clinical features: age of onset, mode of onset | 2 years
  age of onset, mode of onset
The presense of clinical symptoms of patients | 2 years
  The number and severity of clinical symptoms of patients.
Incidence of complications in patients with different treatment regimens | 2 years
  The electronic medical record system was used to collect patients' complications from baseline (admission) to 24 months, and the incidence of complications of different treatment options was compared.
length of hospital stay | 2 years
proportion of patients admitted to ICU | 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Wuhan Pulmonary Hospital(Wuhan Institute for Tuberculosis Control), Hubei, Wuhan